CLINICAL TRIAL: NCT06956131
Title: Metabolite Changes Following Consumption Of Different Protein Drinks In Singapore Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Bezos Earth Fund (Unknown)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: S31; NUS-IRB-2025-19 (Other: National University of Singapore Institutional Review Board (NUS IRB))
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Aging; Protein Metabolism
Keywords: Older adults; Metabolomics; Protein intake; Protein metabolism; Acute; Postprandial; Cognitive function; Mood; Appetite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Casein Protein Drink (Experimental): 30 g protein equivalent of casein protein isolate dissolved in ~250 mL of water
  Interventions: Dietary Supplement: Casein Protein Isolate Drink
- Whey Protein Drink (Experimental): 30 g protein equivalent of whey protein isolate dissolved in ~250 mL of water
  Interventions: Dietary Supplement: Whey Protein Isolate Drink
- Soy Protein Drink (Experimental): 30 g protein equivalent of soy protein isolate dissolved in ~250 mL of water
  Interventions: Dietary Supplement: Soy Protein Isolate Drink
- Maltodextrin Drink (Placebo Comparator): 30 g carbohydrate equivalent of maltodextrin powder dissolved in ~250 mL of water
  Interventions: Dietary Supplement: Maltodextrin Drink

INTERVENTIONS:
Dietary Supplement: Casein Protein Isolate Drink — 30 g protein equivalent of casein protein isolate dissolved in ~250 mL of water
  Arms: Casein Protein Drink
Dietary Supplement: Whey Protein Isolate Drink — 30 g protein equivalent of whey protein isolate dissolved in ~250 mL of water
  Arms: Whey Protein Drink
Dietary Supplement: Soy Protein Isolate Drink — 30 g protein equivalent of soy protein isolate dissolved in ~250 mL of water
  Arms: Soy Protein Drink
Dietary Supplement: Maltodextrin Drink — 30 g carbohydrate equivalent of maltodextrin powder dissolved in ~250 mL of water
  Arms: Maltodextrin Drink

SUMMARY:
The study aims to investigate the acute effects of different protein sources (i.e., casein, whey, soy) on metabolomic profiles (e.g., amino acids in the blood), along with other outcomes such as cognitive function, mood, and appetite. While the study does not directly aim to prevent, prognosticate, diagnose, or alleviate any disease, it may provide insights that could inform dietary recommendations and support disease prevention efforts in older adults.

DETAILED DESCRIPTION:
This study will be a double-blind, randomised, placebo-controlled trial using a crossover study design. 25 older adults (aged 60 to 80) will be recruited and assigned to consume 4 different test drinks in a random order on 4 different visits. This study aims to investigate whether higher protein consumption of different sources will influence postprandial plasma and urinary metabolomic profiles, cognition, mood and appetite. The study will comprise 1 screening visit and 4 test visits separated separated by a minimum washout period of >7 days

ELIGIBILITY:
Inclusion Criteria:

* English-literate and able to give informed consent
* Adults 60 to 80 years old (inclusive)
* (If applicable) Postmenopausal
* BMI of 18·5 to 30 kg/m2 (inclusive)

Exclusion Criteria:

* Currently participating in another clinical study that involves altering the regular diet and/or involves consuming a dietary supplement or investigated food product as an intervention
* Weight change >3 kg in the past 3 months
* Exercising vigorously over the past 3 months (i.e., engaging in high-intensity exercises for more than 3 hours a week, where high-intensity exercises leave one out of breath and unable to talk or sing during the workout)
* Current smokers or have quit smoking for less than 5 years
* Drinking >2 alcoholic drinks per day (i.e., one drink is defined as either 150 ml of wine, 340 ml of beer/cider or 45 ml of distilled spirit)
* If drinking ≤2 alcoholic drinks per day, not willing to stop consumption of alcoholic beverages two days before and on the day of the test visits (total 12 days)
* Not willing to stop consumption of caffeinated beverages 10 to 12 hours before and on the day of the test visits (total 4 days)
* Taking supplements containing omega-3, magnesium, gamma-aminobutyric acid (GABA), L-theanine, melatonin and/or 5-hydroxytryptophan for the past 3 months, and not willing to discontinue usage 3 months before and during the study duration
* Currently on a specialised diet (e.g., vegetarian, vegan, weight loss diet)

  * Had serious food allergies in the past, or having intolerance, sensitivities or allergies to any of the following: milk/dairy products (e.g., casein, whey), starch/starch-derived products (e.g., rice, corn, wheat, potato), soy/soy-derived products, gluten, eggs, nuts, peanuts, fish and crustaceans.
* Disease or impairment of the kidney and/or liver
* Currently diagnosed with diabetes, sleep disorders, gastrointestinal issues (e.g., lactose intolerance, irritable bowel syndrome), gout and/or G6PD deficiency
* History of diseases known to affect the central nervous system (e.g., heart disease, stroke, migraine headaches, multiple sclerosis, Parkinson's disease, mental illnesses)
* Taking antibiotics 2 weeks prior to study participation
* Taking medication known to interfere with cognitive function and mental wellbeing (e.g., benzodiazepines, antidepressants, other central nervous agents)
* Taking anti-hypertensive or cholesterol-lowering drugs for less than 3 years unless medically declared by an official doctor to be in stable condition
* Poor peripheral venous access based on past experiences with blood drawing

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-29 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolites found in plasma (plasma metabolomics) | Baseline, 15, 30, 60, 90, 120, 180, 240, 300 minutes
  Untargeted metabolomics profiling of plasma will be conducted using ultra performance liquid chromatography-quadrupole time of flight-mass spectrometry (UPLC-QTOF-MS)
Changes in metabolites found in urine (urinary metabolomics) | Baseline, 60, 120, 180, 240, 300 minutes
  Untargeted metabolomics profiling of urine will be conducted using ultra performance liquid chromatography-quadrupole time of flight-mass spectrometry (UPLC-QTOF-MS)

SECONDARY OUTCOMES:
Cognitive Function | Baseline, 15, 60, 120, 180, 240, 300 minutes
  The Computerised Mental Performance Assessment System (COMPASS) will be administered via a laptop. The COMPASS tests consist of 5 consecutive tests, including Digit Vigilance, Stroop, Rapid Visual Information Processing, Computerised Corsi Blocks Lite, Alphabetic Working Memory and Serial Subtraction, where the correctness and reaction time will be recorded. The test is expected to take around 15 minutes.
Mood | Baseline, 15, 60, 120, 180, 240, 300 minutes
  The Profile of Mood States (POMS) questionnaire will be administered, which contains various words that describe feelings. Participants will indicate, for each word, how they currently feel on scale of 0 (Not at all) to 4 (Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Ph.D., R.D., Principal Investigator — National University of Singapore, Department of Food Science and Technology
Locations (1):
- NUS, Department of Food Science and Technology, 1 Science Drive 3, Block S13, #03-07, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on NUS OneDrive with access limited only Dr Kim Jung Eun and her research staff. All data will be de-identified prior to statistical analyses.

REFERENCES:
- [Background] Lanng SK, Oxfeldt M, Johansen FT, Risikesan J, Hansen M, Bertram HC. Acute changes in the metabolome following resistance exercise combined with intake of different protein sources (cricket, pea, whey). Metabolomics. 2023 Nov 24;19(12):98. doi: 10.1007/s11306-023-02064-0. PMID 37999866